CLINICAL TRIAL: NCT05176340
Title: Effect of Action Modules on Resilience and Psychological Health of Stroke Patients
Brief Title: Action Modules on Resilience and Psychological Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Hsiang Chu Pai, Principal Investigator, Chung Shan Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CS2-18011
Record Dates: First submitted 2021-12-04; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Stroke Patients
Keywords: anxiety; depression; resilience; illness representation
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The Specific Thematic Nursing Care Action Modules (STNC-AM) platform that we present here is an educational program that integrates education and coaching. STNC-AM has six key aspects: stroke prevention, management of emotions, management of fatigue, physical activity, caregiver training, and integrative resources. Each scope contains detailed care guidance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the experimental group were provided an education program through the Care Action Module during their hospitalization period, and follow-up was conducted one and two months after discharge.
  Interventions: Other: Specific Thematic Nursing Care Action Modules (STNC-AM)
- Control group (No Intervention): The control group received no intervention, except for the regular care followed by the nurses in general in the rehabilitation ward.

INTERVENTIONS:
Other: Specific Thematic Nursing Care Action Modules (STNC-AM) — The STNC-AM platform that investigators present here is an educational program that integrates education and coaching.
  The nurse coaching component was based on the STNC-AM platform. This online platform can guide nurses' health education for the comprehensive care of stroke patients. Nurses can use an iPad and enter the STNC-AM platform website, where they can directly access the Care Action Module.
  Arms: Intervention group

SUMMARY:
This study aimed to determine whether interventions that use the Specific Thematic Nursing Care Action Modules (STNC-AM) platform improve patients' psychological health over a two-month period.

DETAILED DESCRIPTION:
The STNC-AM platform that investigator present here is an educational program that integrates education and coaching. STNC-AM has six key aspects: stroke prevention, management of emotions, management of fatigue, physical activity, caregiver training, and integrative resources. Each scope contains detailed care guidance. The nurse coaching component was based on the six key aspects detailed above. This online platform can guide nurses' health education for the comprehensive care of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* remaining hospitalized within 6 months after a stroke attack.
* being able to communicate verbally.
* being willing to participate.

Exclusion Criteria:

* Aphasia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Illness Perception_change is being assessed | The data collection was conducted at three time points: first week (baseline; Time 1) of admission to the rehabilitation ward and then first month (Time 2) and second month (Time 3) follow-up after discharge.
  Investigators used the Illness Perception Questionnaire-Revised (IPQ-R) to evaluate stroke patients' positive illness representation.
  Investigators used the three positive domains (personal control, treatment control, and illness coherence) of illness representation to evaluate stroke patients' positive illness representation. Total scores ranged from 16 to 80 in each domain. High scores on all three dimensions (personal control, treatment control, and illness coherence) indicated a more positive illness representation.
Depression and Anxiety_change is being assessed | The data collection was conducted at three time points: first week (baseline; Time 1) of admission to the rehabilitation ward and then first month (Time 2) and second month (Time 3) follow-up after discharge.
  Investigators used the Hospital Anxiety and Depression Scale (HADS) to evaluate stroke patients' depression and anxiety.Total scores ranged from 0 to 21 in each domain, and higher scores indicated higher anxiety or depression.
Resilience_change is being assessed | The data collection was conducted at three time points: first week (baseline; Time 1) of admission to the rehabilitation ward and then first month (Time 2) and second month (Time 3) follow-up after discharge.
  Investigators used the Resilience Scale (RS) to evaluate stroke patients' resilience.Total scores ranged from 25 to 175, with higher scores as indicating greater resilience

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan